CLINICAL TRIAL: NCT00610610
Title: Paroxetine-CR (Paxil-CR) in the Treatment of Patients With Fibromyalgia Syndrome: A Randomized, Double Blind, Parallel Group, Flexible Dose, Placebo Controlled Trial.
Brief Title: Paroxetine-CR (Paxil-CR) in the Treatment of Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Ashwin A Patkar / M.D, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3610; IRB#3610
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2008-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; Paroxetine
MeSH Terms: conditions — Fibromyalgia | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Paroxetine - Controlled Release
  Interventions: Drug: Paroxetine CR
- B (Placebo Comparator): Same colour, shape placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine CR — Those in the active treatment group will receive doses of Paxil CR in the following manner: week 1: 12.5 mg per day, week 2: 25 mg per day, week 3: 37.5 mg per day, wk 4: 50 mg per day and week 5: 62.5 mg per day.
  Other Names: Paxil CR
  Arms: A
Drug: Placebo — Same shape Placebo
  Arms: B

SUMMARY:
Objective: Although there is a high comorbidity of depressive and/or anxiety disorders with fibromyalgia, information on the clinical implications of this comorbidity is limited. We investigated whether a history of depressive and/or anxiety disorders was associated with response to treatment in a double blind, randomized, placebo controlled trial of paroxetine controlled release (CR) in fibromyalgia.

Method: One hundred and sixteen fibromyalgia subjects were randomized to receive paroxetine CR (dose 12.5-62.5 mg/day) or placebo for 12 weeks. The Mini International Neuropsychiatric Interview (M.I.N.I-plus) was used to ascertain current or past diagnoses of depressive and anxiety disorders. Patients with current depressive or anxiety disorders were excluded, but those with past diagnoses were enrolled in the trial. Subjective depression and anxiety were assessed using the Beck Depression Inventory (BDI) and the Beck Anxiety Inventory (BAI); subjects were excluded if they scored greater than 23 on the BDI. Health Status was determined using the 36-Item Short Form Health Survey (SF-36), the Sheehan Disability Scale (SDS), the Perceived Stress Scale (PSS) and the Pittsburgh Sleep Quality Index (PSQI). The primary outcome was treatment response defined as ≥ 25% reduction in the Fibromyalgia Impact Questionnaire (FIQ) score. Secondary outcomes included changes in scores on the Clinical Global Impression-Severity and Improvement (CGI-S and CGI-I respectively), the Visual Analogue Scale for Pain (VAS) scores and number of tender points.

DETAILED DESCRIPTION:
Introduction

Despite the skepticism of some physicians over the very existence of a condition called Fibromyalgia syndrome (FMS), most agree that this is a common condition seen in pain clinics. The syndrome is characterized by widespread pain (1) persistent fatigue (2), and non restorative sleep (3), and generalized morning stiffness (4). Other syndromes are also frequently seen and include headaches, TMJ, irritable bowel syndrome, depression, anxiety, paresthesias and memory loss. FMS may be primary or secondary to other disease states. Conditions like hypothyroidism may mimic FMS. The prevalence of depression is about 30-35% (1). FMS affects more women than men (20:1) and the prevalence increases with age so that about 7% of women over 70 years of age are affected compared to the prevalence rate of about 2% in the general population.

The diagnosis is based on patients complaints of pain and a clinical examination of multiple tender points (11/18) as defined by the ACR criteria for FMS (8) or (11 or less) per Copenhagen declaration. There is no specific laboratory test for FMS.

The causes are unknown, but many investigators believe that FMS encompasses a spectrum of diseases with a common pathogenic pathway. Links between FMS and non-restorative deep sleep has been reported (2). Other changes frequently seen in FMS patients include elevated interleukin-2 (3), low levels of serum serotonin and its precursor tryptophan (4) and elevated substance -P levels (5). There has been increasing interest in the effect of serotonin on pain in recent years. Serum serotonin levels have been shown to be significantly lower in fibromyalgia patients than in those without fibromyalgia (6). Evidence is available to suggest that administration of the serotonin precursor tryptophan improves pain symptoms in a variety of patient cohorts. (7)

Treatment is generally multidisciplinary with an emphasis on active patient participation, cognitive behavioral therapy, physical modalities and medications. (9). A review of the literature reveals that there is no consensus for the pharmacological treatment for FMS. A rational polypharmacy is advocated with medications used to improve pain, sleep, fatigue and other associated symptoms. (10) Oral agents utilized for symptomatic relief include acetaminophen, non-steroidal anti-inflammatory medications, and steroids. Each is associated with potentially serious medical sequelae with chronic use, and results have been disappointing. Cyclobenzaprine (flexeril) has shown efficacy for FMS though common side effects, such as dry mouth and drowsiness, can limit its use. (11) Benzodiazepines and opiates, which are also utilized for FMS are potentially addictive. Modafinil (Provigil) has been used to treat the fatigue associated with FMS (12). Case reports have indicated the usefulness of atypical antipsychotics like olanzapine for the treatment of FMS symptoms (13). No one medication has been found to control all the symptoms of FMS and the goal of therapy is to improve pain, function and quality of life by combining the least amount of medications.

There have been 21 controlled trials involving antidepressants, most involving tricyclic antidepressants. A recent meta analysis revealed that compared to placebo, the effect sizes for tricyclic antidepressants were substantially larger than zero for all measurements (14). Two randomized placebo controlled trials have examined the SSRI fluoxetine (20 mg per day for 6 weeks) (15,16) and two have examined the SSRI citalopram (20-40 mg per day for 8 weeks) (17, 18) in the treatment of FMS. These studies had equivocal results; but the trials were limited by a high dropout rate in the placebo group, a brief trial duration and small sample sizes.

In a more recent study, Wetherhold et al, examined 82 women with fibromyalgia, randomized to receive either paroxetine (20 mg/day), nabumetone (2000 mg/day) or a combination of paroxetine (20 mg/day) and nabumetone (2000 mg/day). Patient received each treatment regimen for a period of 8 weeks. The study demonstrated that the combination regimen was superior to nabumetone alone, but not to paroxetine alone, in improving the signs and symptoms of fibromyalgia - suggesting that paroxetine was responsible for the improvement in the combined regimen (19).

Thus, a non-addictive oral agent, with dual action (NE and 5 HT reuptake blockade) and a relatively benign side effect profile such as paroxetine (Paxil), has the potential to be a significant addition to the treatment of FMS. Moreover, paroxetine's side effect profile is favorable to tricyclic antidepressants and therefore would likely be a preferable treatment option if effective. A recent extended release preparation of paroxetine (Paxil CR) is prudentially absorbed in the intestine rather than the stomach and is reported to have a more favorable GI side effect profile and may be particularly suitable for the study. The agent could be used alone or adjunctively to decrease the patient's requirement for other analgesic medications.

This study proposes to study Paxil CR, a selective serotonin reuptake inhibitor, to treat FMS with particular emphasis on its effect on the full constellation of symptoms associated with this disorder and quality of life improvement in this patient population.

In our experience physicians from multiple specialties (family medicine/neurology/physiatry/rheumatology/pain medicine/psychiatry) are increasingly discussing anecdotal reports of the efficacy of SSRIs in treating FMS symptoms. This study protocol is intended to evaluate the efficacy of this practice. It is our hypothesis that paroxetine will be shown to be an effective addition to the treatment as defined below.

Study Design:

Randomized, double blind, parallel group, flexible dose, placebo controlled 12-week study.

Subject number: One hundred and twenty five.

Study Schedule: (see attached schedule of evaluations)

Patients will be screened for eligibility based on a confirmed diagnosis of FMS (per report of rheumatologist or treating specialist). Only those meeting eligibility criteria (inclusion/exclusion criteria) will be permitted to give informed consent to enter the study. Psychological assessments will be performed using standardized questionnaires at screening, baseline and defined time points in the study as described in the schedule of evaluations. After a blood draw for routine labs to exclude other potential treatable conditions, and pregnancy test (for women), urine testing for illicit drugs and EKG, the participants will enter a one- week placebo lead-in period; those that show a less than 25% reduction on FIQ will enter the randomization phase. The routine labs will include the CBC with differential, SMA-7, liver function tests, thyroid panel, Anti Nuclear antibody (ANA), Rheumatoid factor (Rh factor), Anti Polymerase Antibody (APA), C-Reactive protein and Erythrocyte Sedimentation Rate (ESR). Patients will be instructed to swallow the tablets whole and not to crush or chew them via labels on the medication bottles. Eligible study participants will be randomized to either paroxetine or placebo (60 patients in each arm). Those in the active treatment group will receive doses of Paxil CR in the following manner: week 1: 12.5 mg per day, week 2: 25 mg per day, week 3: 37.5 mg per day, wk 4: 50 mg per day and week 5: 62.5 mg per day. Patients who do not tolerate higher doses will be maintained on the minimum tolerated dose. The placebo arm will be treated identically except for the content of the capsules. The total duration of active treatment will be 12 weeks. Patients will be seen weekly for the first 4 weeks and biweekly thereafter. After the final visit, the study medication will be tapered over 2 weeks.

Unblinding procedures in case of emergency:

A list of patient randomization numbers and corresponding treatments will be available with local Pharmacy. In case of emergency local pharmacy can be called (24 hours) to reveal the study assignment of the patients. Once blind is broken, the patient will be immediately discontinued from the study but will be evaluated and treated as warranted by their clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia according to American College of Rheumatology criteria
* A pain score of > 5 cm on a 0 to 10 Visual Analogue Scale
* < 23 on the Beck Depression Inventory-II.
* 18 and 65 years of age
* Ability to give informed consent
* If patients are of child-bearing potential, an effective contraceptive was required (i.e., oral, depo-provera, or implanted contraceptives, an IUD, a diaphragm or condom with spermicide or abstinence) for at least one month prior to the Screening Visit and have a negative pregnancy test upon entry into the study.

Exclusion Criteria:

* Diagnosis of systemic lupus erythematous or other connective tissue disorders (e.g., scleroderma, polymyositis, sjogren's syndrome).
* Diagnosis of myopathy, muscular dystrophy, rheumatoid arthritis, crystal induced arthritis.
* Involvement in a litigation concerning fibromyalgia or silicone breast implant disease
* Use of antidepressant medications (including MAO Inhibitors) within the previous week or previous 5 weeks for fluoxetine.
* History of allergy or hypersensitivity to NSAIDs or antidepressants.
* Treatment with an investigational drug within 30 days prior to the Screening Visit.
* Treatment with corticosteroids within 14 days prior to the Screening Visit or acupuncture treatment within 21 days prior to the Screening Visit.
* Analgesic and sedative medication doses will remain unchanged during the treatment.
* Patients on antidepressants for mood and anxiety disorders.
* Current or previous history of bipolar disorder, schizophrenia, schizoaffective disorder or major somatization disorder.
* Current diagnosis of major depression or anxiety disorder on the MINI.
* Hospitalization for psychotic episode or attempted suicide within one year of study entry.
* Current substance abuse or history of substance abuse in the previous 12 months.
* Diagnosis of uncontrolled hypothyroidism or brittle diabetes.
* History of bleeding diathesis of any etiology.
* History of chronic hepatitis or cirrhosis.
* Glaucoma
* Presence of active gastrointestinal bleeding or an active ulcer within one month prior to the Screening Visit.
* Significant cardiac, pulmonary, metabolic, renal, or hepatic disease, or history of malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Twenty five percent change from baseline in Fibromyalgia Impact Questionnaire (FIQ) total scores | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in FIQ, Number of tender points, Beck Depression Inventory II, Beck Anxiety Inventory, Visual Analog Scale for pain | 12 weeks
Recording of spontaneous adverse events throughout the screening, run-in, and treatment phases of the study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin A Patkar, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania